CLINICAL TRIAL: NCT03445845
Title: Rotation or Change of Biotherapy After TNF Blocker Treatment Failure for Axial Spondyloarthritis
Acronym: ROC-SPA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1608185; 2017-004700-22 (EudraCT Number)
Record Dates: First submitted 2018-02-20; First posted 2018-02-26 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Axial Spondyloarthritis
Keywords: TNF blocker; change of biotherapy
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — secukinumab; Tumor Necrosis Factor Inhibitors; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- targeting IL-23/17 axis (Experimental): The experimental group (targeting IL-23/17 axis) receiving secukinumab in compliance with the marketing authorization regimen: 150 mg per week for 5 weeks, and then every month by subcutaneous injection.
  Blood specimen at each visits
  Interventions: Drug: Secukinumab; Biological: blood specimen
- TNF blocker (Active Comparator): • The control group receiving a second TNF blocker in compliance with the marketing authorization regimen:
  The TNF blocker (originator or biosimilar) will be different to the TNF used before the inclusion and will be chose by the investigator:
  * infliximab: 5mg/kg per IV infusion at weeks 0, 2, 6, and then every 6 weeks,
  * etanercept: 50mg per week in subcutaneous injection,
  * adalimumab: 40mg every other week in subcutaneous injection,
  * certolizumab: 400mg every other week 3 times, and then 200mg every other week or 400mg per month in subcutaneous injections,
  * golimumab: 50mg every month in subcutaneous injection, in case of overweight (>100kg) an inadequate response, 100mg every month is allow.
  Blood specimen at each visits
  Interventions: Drug: TNF blocker; Biological: blood specimen

INTERVENTIONS:
Drug: Secukinumab — Secukinumab : 150 mg per week for 5 weeks, and then every month by subcutaneous injection
  Arms: targeting IL-23/17 axis
Drug: TNF blocker — TNF blocker (originator or biosimilar) :
  * infliximab: 5mg/kg per IV infusion at weeks 0, 2, 6, and then every 6 weeks,
  * etanercept: 50mg per week in subcutaneous injection,
  * adalimumab: 40mg every other week in subcutaneous injection,
  * certolizumab: 400mg every other week 3 times, and then 200mg every other week or 400mg per month in subcutaneous injections,
  * golimumab: 50mg every month in subcutaneous injection, in case of overweight (>100kg) an inadequate response, 100mg every month is allow.
  Arms: TNF blocker
Biological: blood specimen — Blood specimen at each visits for measurement of bDMARS blockers concentration and anti-drug antibody concentration

SUMMARY:
Axial spondyloarthritis (axSpA) is a chronic inflammatory disease characterized by inflammatory arthritis and enthesitis involving the spine. AxSpA prevalence is around 0.17% of the French population. Tumor necrosis factor (TNF) was the first target defined in axSpA. Since one third of axSpA patients failed to the first TNF blocker, many axSpA patients received a second biological Disease-Modifying AntiRheumatic Drugs (bDMARDs). Until few months, the only choice was to use a second TNF blocker.Since 2003, pharmaceutical companies investigated efficacy of TNF blockers already used in rheumatoid arthritis. Etanercept is a fusion protein with TNF receptor type II p75 and IgG1 Fc fragment, whereas adalimumab, infliximab, and golimumab are monoclonal antibodies. Certolizumab is a fusion between a fab fragment targeting TNF and a Peg fraction. All demonstrated efficacy versus placebo in a randomized double blinded study

In case of failure to the first TNF blockers, rheumatologists will follow the "Treat-to-Target" principle. This approach already demonstrated its benefit in rheumatoid arthritis or in psoriatic arthritis. This concept was also suggested for axSpA with low levels of evidence and recommendation. So rheumatologist will provide the best treatment in case of failure to the first TNF blockers, which is a daily clinical situation. Since few months, rheumatologists have the choice between targeting IL-23/17 axis compared to a second TNF blocker.

ELIGIBILITY:
Inclusion Criteria:

* Active axSPA with BASDAI>4 or ASDAS>3.5, who need change in TNF blocker treatment
* Aged over 18 years
* Inadequate response after at least 3 months to the 1st TNF blocker
* If non biologic DMARD treatment : stable dose for at least on month before inclusion
* If oral corticosteroids treatment : stable dose for at least on month before inclusion
* If NSAIDs treatment : stable dose for at least on month before inclusion
* Ability to complete questionnaires
* Social security affiliation
* Informed written consent given

Exclusion Criteria:

* Any contra-indication to TNF blocker and/or secukinumab
* Inflammatory bowel diseases
* Existing pregnancy, lactation, or intended pregnancy within the next 15 months Active tuberculosis or other severe infections such as sepsis or opportunistic infections
* Active infections, including chronic or localised infections.
* Moderate to severe heart failure (NYHA classes III/IV)
* Impossibility to give informed consent
* Impossibility to be followed for 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2024-09-21 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Proportion of axSpA patients with a clinical response Assessments in Ankylosing Spondylitis International Society 40 (ASAS 40) at week 24 | 24 weks
  ASAS 40 is defined as an improvement of at least 40% and absolute improvement of at least 2 units on a numerical rating scale of 10 in at least 3 of the following domains compared to values at inclusion:
  * Patient global assessment : numerical rating scale with extremes labelled "none" and "severe."
  * Pain assessment : average of total and nocturnal pain scores, both measured on a numerical rating scale with extremes labelled "no pain" and "most severe pain."
  * Function : BASFI average of 10 questions measured by numerical rating scale with extremes labelled "easy" and "impossible."
  * Morning stiffness, represented by the average of the last 2 questions on the 6-question BASDAI measured by numerical rating scale: one with extremes labelled "none" and "very severe"; the other marking duration of morning stiffness between "0" and "2 or more hours." Additionally, no worsening at all in remaining domain

SECONDARY OUTCOMES:
Proportion of axSpA patients with a clinical response ASAS 40 at week 12 | 12 weeks
  ASAS 40 is defined as an improvement of at least 40% and absolute improvement of at least 2 units on a numerical rating scale of 10 in at least 3 of the following domains compared to values at inclusion:
  * Patient global assessment : numerical rating scale with extremes labelled "none" and "severe."
  * Pain assessment : average of total and nocturnal pain scores, both measured on a numerical rating scale with extremes labelled "no pain" and "most severe pain."
  * Function : BASFI average of 10 questions measured by numerical rating scale with extremes labelled "easy" and "impossible."
  * Morning stiffness, represented by the average of the last 2 questions on the 6-question BASDAI measured by numerical rating scale: one with extremes labelled "none" and "very severe"; the other marking duration of morning stiffness between "0" and "2 or more hours." Additionally, no worsening at all in remaining domain
Proportion of axSpA patients with a clinical response ASAS 40 at week 52 | 52 weeks
  ASAS 40 is defined as an improvement of at least 40% and absolute improvement of at least 2 units on a numerical rating scale of 10 in at least 3 of the following domains compared to values at inclusion:
  * Patient global assessment : numerical rating scale with extremes labelled "none" and "severe."
  * Pain assessment : average of total and nocturnal pain scores, both measured on a numerical rating scale with extremes labelled "no pain" and "most severe pain."
  * Function : BASFI average of 10 questions measured by numerical rating scale with extremes labelled "easy" and "impossible."
  * Morning stiffness, represented by the average of the last 2 questions on the 6-question BASDAI measured by numerical rating scale: one with extremes labelled "none" and "very severe"; the other marking duration of morning stiffness between "0" and "2 or more hours." Additionally, no worsening at all in remaining domain
Proportion of axSpA patients with a clinical response ASAS 20 at week 12 | 52 weeks
  ASAS 20 is defined as an improvement of at least 20% and absolute improvement of at least 1 unit on a numerical rating scale of 10 in at least 3 of the following domains compared to values at inclusion:
  * Patient global assessment : numerical rating scale with extremes labelled "none" and "severe."
  * Pain assessment : average of total and nocturnal pain scores, both measured on a numerical rating scale with extremes labelled "no pain" and "most severe pain."
  * Function : BASFI average of 10 questions regarding measured by numerical rating scale with extremes labelled "easy" and "impossible."
  * Morning stiffness, represented by the average of the last 2 questions on the 6-question BASDAI measured by numerical rating scale: one with extremes labelled "none" and "very severe"; the other marking duration of morning stiffness between "0" and "2 or more hours." Additionally, no worsening in a similar amount in the fourth domain
Proportion of axSpA patients with a clinical response ASAS 20 at week 24 | 24 weeks
  ASAS 20 is defined as an improvement of at least 20% and absolute improvement of at least 1 unit on a numerical rating scale of 10 in at least 3 of the following domains compared to values at inclusion:
  * Patient global assessment : numerical rating scale with extremes labelled "none" and "severe."
  * Pain assessment : average of total and nocturnal pain scores, both measured on a numerical rating scale with extremes labelled "no pain" and "most severe pain."
  * Function : BASFI average of 10 questions regarding measured by numerical rating scale with extremes labelled "easy" and "impossible."
  * Morning stiffness, represented by the average of the last 2 questions on the 6-question BASDAI measured by numerical rating scale: one with extremes labelled "none" and "very severe"; the other marking duration of morning stiffness between "0" and "2 or more hours." Additionally, no worsening in a similar amount in the fourth domain
Proportion of axSpA patients with a clinical response ASAS20 at week 52 | 52 weeks
  ASAS 20 is defined as an improvement of at least 20% and absolute improvement of at least 1 unit on a numerical rating scale of 10 in at least 3 of the following domains compared to values at inclusion:
  * Patient global assessment : numerical rating scale with extremes labelled "none" and "severe."
  * Pain assessment : average of total and nocturnal pain scores, both measured on a numerical rating scale with extremes labelled "no pain" and "most severe pain."
  * Function : BASFI average of 10 questions regarding measured by numerical rating scale with extremes labelled "easy" and "impossible."
  * Morning stiffness, represented by the average of the last 2 questions on the 6-question BASDAI measured by numerical rating scale: one with extremes labelled "none" and "very severe"; the other marking duration of morning stiffness between "0" and "2 or more hours." Additionally, no worsening in a similar amount in the fourth domain
Proportion of axSpA patients with a partial remission rate at week 12 | 12 weeks
  Partial remission is defined by values lower than 2/10 in each 4 domains:
  * Patient global assessment measured on a numerical rating scale with extremes labelled "none" and "severe."
  * Pain assessment represented by the average of total and nocturnal pain scores, both measured on a numerical rating scale with extremes labelled "no pain" and "most severe pain."
  * Function represented by BASFI average of 10 questions regarding ability to perform specific tasks as measured by numerical rating scale with extremes labelled "easy" and "impossible."
  * Morning stiffness, represented by the average of the last 2 questions on the 6-question BASDAI regarding morning stiffness as measured by numerical rating scale: one with extremes labelled "none" and "very severe"; the other marking duration of morning stiffness between "0" and "2 or more hours."
Proportion of axSpA patients with a partial remission rate at week 24 | 24 weeks
  Partial remission is defined by values lower than 2/10 in each 4 domains:
  * Patient global assessment measured on a numerical rating scale with extremes labelled "none" and "severe."
  * Pain assessment represented by the average of total and nocturnal pain scores, both measured on a numerical rating scale with extremes labelled "no pain" and "most severe pain."
  * Function represented by BASFI average of 10 questions regarding ability to perform specific tasks as measured by numerical rating scale with extremes labelled "easy" and "impossible."
  * Morning stiffness, represented by the average of the last 2 questions on the 6-question BASDAI regarding morning stiffness as measured by numerical rating scale: one with extremes labelled "none" and "very severe"; the other marking duration of morning stiffness between "0" and "2 or more hours."
Proportion of axSpA patients with a partial remission rate at week 52 | 52 weeks
  Partial remission is defined by values lower than 2/10 in each 4 domains:
  * Patient global assessment measured on a numerical rating scale with extremes labelled "none" and "severe."
  * Pain assessment represented by the average of total and nocturnal pain scores, both measured on a numerical rating scale with extremes labelled "no pain" and "most severe pain."
  * Function represented by BASFI average of 10 questions regarding ability to perform specific tasks as measured by numerical rating scale with extremes labelled "easy" and "impossible."
  * Morning stiffness, represented by the average of the last 2 questions on the 6-question BASDAI regarding morning stiffness as measured by numerical rating scale: one with extremes labelled "none" and "very severe"; the other marking duration of morning stiffness between "0" and "2 or more hours."
Proportion of axSpA patients with a ASDAS major improvement at week 12 | 12 weeks
  ASDAS major improvement was defined by a variation of ASDAS-CRP≥2
Proportion of axSpA patients with a ASDAS major improvement at week 24 | 24 weeks
  ASDAS major improvement was defined by a variation of ASDAS-CRP≥2
Proportion of axSpA patients with a ASDAS major improvement at week 52 | 52 weeks
  ASDAS major improvement was defined by a variation of ASDAS-CRP≥2
Proportion of axSpA patients with biological Disease-Modifying AntiRheumatic Drugs (bDMARDs) treatment at week 12 | 12 weeks
  Patient with the same bDAMRs treatment at inclusion and week 12
Proportion of axSpA patients with biological Disease-Modifying AntiRheumatic Drugs (bDMARDs) treatment at week 24 | 24 weeks
  Patient with the same biological Disease-Modifying AntiRheumatic Drug (bDAMR) treatment at inclusion and week 24
Proportion of axSpA patients with bDMARDs treatment at week 52 | 52 weeks
  Patient with the same biological Disease-Modifying AntiRheumatic Drug (bDAMR) treatment at inclusion and week 52
Number of adverse events | 52 weeks
  Number of adverse events
Correlation between concentration of antibodies to bDMARS blockers and clinical response according to treatment | From baseline to 52 weeks
  Concentration of antibodies to bDMARS blockers is measured by Enzyme Linked ImmunoSorbent Assay (ELISA) low disease activity is defined by BASDAI <4 and ASDAS <2.1
Correlation between concentration of anti-drug antibodies and clinical response according to treatment | From baseline to 52 weeks
  Concentration of anti-drug antibodies is measured by Enzyme Linked ImmunoSorbent Assay (ELISA) low disease activity is defined by BASDAI <4 and ASDAS <2.1

CONTACTS AND LOCATIONS:
Overall Officials: Hubert MAROTTE, MD, Study Director — CHU SAINT-ETIENNE
Locations (35):
- France (34):
  - CHU d'Angers, Angers
  - CHRU Besançon, Besançon
  - APHP- Hôpital Avicenne, Bobigny
  - CHU Bordeaux, Bordeau
  - CHRU Brest, Brest
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU de Grenoble Alpes, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - CH Le Mans, Le Mans
  - CHRU Lille, Lille
  - Hôpital Saint-Philibert, Lomme
  - CH Lyon SUD, Lyon
  - Hôpital Edouard Herriot, Lyon
  - CHRU Montpellier, Montpellier
  - CHU Montpellier - 2 - Unité Clinique thérapeutique des Maladies Ostéo-Articulaires, Montpellier
  - CHU Nancy, Nancy
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - CHR d'Orléans, Orléans
  - APHP - Hôpital Ambroise Paré, Paris
  - APHP - Hôpital Bichat, Paris
  - APHP - Hôpital Cochin, Paris
  - APHP - Hôpital Henri Mondor, Paris
  - APHP - Hôpital Lariboisière, Paris
  - APHP - Hôpital Pitié-Salpétrière, Paris
  - APHP - Hôpital Saint-Antoine, Paris
  - APHP - Kremlin-Bicêtre, Paris
  - CHU de Poitiers, Poitiers
  - CHU Reims, Reims
  - CHU de Rouen, Rouen
  - CHU Saint-Etienne, Saint-Etienne
  - CHU STRASBOURG - Hautepierre, Strasbourg
  - CHU Toulouse, Toulouse
  - CHRU Tours, Tours
- CH Princesse de Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dalix E, Marcelli C, Bejan-Angoulvant T, Finckh A, Rancon F, Akrour M, De Araujo L, Presles E, Marotte H; ROC-SpA study group. Rotation or change of biotherapy after TNF blocker treatment failure for axial spondyloarthritis: the ROC-SpA study, a randomised controlled study protocol. BMJ Open. 2024 Sep 10;14(9):e087872. doi: 10.1136/bmjopen-2024-087872. PMID 39260856